CLINICAL TRIAL: NCT00005856
Title: Phase I/II Trial of Oxaliplatin as Neoadjuvant Treatment in Adults With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Oxaliplatin in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02336; 9902; U01CA062475 (NIH); CDR0000067883 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Oxaliplatin

ARMS (1):
- Treatment (oxaliplatin) (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: oxaliplatin; Other: pharmacological study

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of oxaliplatin in treating patients with newly diagnosed glioblastoma multiforme. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of oxaliplatin in patients with newly diagnosed glioblastoma multiforme who are receiving or not receiving anticonvulsants known to be metabolized by P450.

II. Determine the dose-limiting toxicity and safety profile of this drug in this patient population.

III. Assess the pharmacokinetics of this drug on this schedule and determine the effects of P450-inducing anticonvulsants on the pharmacokinetics in these patients.

IV. Determine the radiographic response rate in patients treated with this drug.

V. Determine survival and drug toxicity in these patients.

OUTLINE: This is a phase I dose-escalation study of oxaliplatin followed by a phase II study. Patients are stratified according to whether concurrent anticonvulsant drugs induce P450 (yes vs modest/no or no drugs).

Phase I: Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients (per stratum) receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Phase II: Patients receive oxaliplatin as in phase I at the MTD determined in phase I.

Patients are followed at 1 month, every 2 months until disease progression, and then monthly thereafter.

PROJECTED ACCRUAL: Approximately 24 patients (12 per stratum) will be accrued for the phase I part of this study within 8-12 months. A total of 18-35 patients will be accrued for the phase II part of this study within 5-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed supratentorial grade IV astrocytoma

  * Glioblastoma multiforme
* Subtotal resection or biopsy with measurable and contrast-enhancing disease on the postoperative, pretreatment MRI/CT scan
* Performance status - Karnofsky 60-100%
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* Bilirubin normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious concurrent infection or medical illness that would jeopardize ability to receive protocol chemotherapy with reasonable safety
* No other prior malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer
* No grade 2 or greater pre-existing sensory neuropathy
* No history of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol chemotherapy
* Mini mental score at least 15
* No prior immunotherapy for glioblastoma multiforme
* No prior biologic therapy for glioblastoma multiforme, including:

  * Immunotoxins
  * Immunoconjugates
  * Antiangiogenesis compounds
  * Antisense
  * Peptide receptor antagonists
  * Interferons
  * Interleukins
  * Tumor infiltrating lymphocytes
  * Lymphokine activated killer cells
  * Gene therapy
* No concurrent filgrastim (G-CSF)
* No prior chemotherapy for glioblastoma multiforme
* No prior hormonal therapy for glioblastoma multiforme
* Prior glucocorticoid therapy for glioblastoma multiforme allowed
* Must be maintained on a stable (lowest required dose) corticosteroid regimen for at least 5 days before and during study
* No concurrent dexamethasone as an antiemetic
* No prior radiotherapy for glioblastoma multiforme
* Recovered from immediate postoperative period
* At least 10 days since prior anticonvulsant drug that induces hepatic metabolic enzymes
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2000-12; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) defined as the dose level at which 2 out of 6 or the dose level below that at which >= 2 of 3 or > 2 of 6 patients experience dose-limiting toxicity (DLT) assessed by Common Toxicity Criteria (CTC) version 2.0 (Phase I) | 14 days
DLT is defined as grade 3 or 4 nonhematological toxicities or hematological toxicities as assessed by CTC version 2.0 (Phase I) | 14 days
Pharmacokinetics of oxaliplatin (Phase I) | At baseline, at immediately post infusion, at 2, 4, 22, and 24 hours (of course 1)

SECONDARY OUTCOMES:
Response rate (Phase II) | Up to 7 years
Duration of survival (Phase II) | Up to 7 years
  Estimated with 95% confidence intervals.
Frequency of toxicity as assessed by CTC version 2.0 (Phase II) | Up to 7 years after completion of study treatment
  The proportion of patients with serious or life threatening toxicities will be estimated along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, Principal Investigator — New Approaches to Brain Tumor Therapy Consortium
Locations (1):
- New Approaches to Brain Tumor Therapy Consortium, Baltimore, Maryland, United States